CLINICAL TRIAL: NCT05710042
Title: Clinical Study of the BioVentrix Revivent TC™ System for Treatment of Left Ventricular Aneurysms ALIVE-EA (American Less Invasive Ventricular Enhancement-Expanded Access)
Brief Title: ALIVE Expended Access - Clinical Study
Acronym: ALIVE-EA
Status: No longer available | Type: Expanded Access
Sponsor: BioVentrix (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-0067
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Left Ventricle Remodeling
Keywords: Heart Failure; Left Ventricular Remodeling
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling

INTERVENTIONS:
Device: Revivent TC System — The Revivent TC System is indicated for patients suffering from symptomatic heart failure referred for treatment of left ventricular antero-septal aneurysms/scars that are contiguous and includes both anterior and septal components.

SUMMARY:
A prospective, multi-center, single-arm study. This study will enroll a maximum of 35 subjects treated with the Revivent TC System.

DETAILED DESCRIPTION:
The purpose of this study is to allow the continued use of the BioVentrix Revivent TC System for the treatment of LV antero-septal aneurysms/scars in patients with symptomatic heart failure while the pivotal trial for the BioVentrix Revivent TC System is continuing through the follow up phase and the PMA documentation is prepared and reviewed by FDA.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older;
2. LV Aneurysm or Scar Presence: Defined by presence of a contiguous acontractile (akinetic and/or dyskinetic) scar;
3. LV Aneurysm/Scar Location: Defined as a scar involving septum and/or anterior, apical or anterolateral regions of the left ventricle as evidenced by cardiac imaging and referred for surgical management;
4. Viability of myocardium in regions remote from area of intended scar exclusion as evidenced by cardiac imaging;
5. Left Ventricular Ejection Fraction < 45%;
6. Left ventricular end-systolic volume index ≥50 mL/m2;
7. Suffering from heart failure symptoms as defined by NYHA Classification > 2 not responsive to medical therapy;
8. Patient completed 6 Minute Walk Test and MLHF Quality of Life Questionnaire (can be performed at baseline visit);
9. Patient is on adequate Guideline Directed Medical Therapy (GDMT);
10. Subject or a legally authorized representative must provide written informed consent;
11. Agree to required follow-up visits; and
12. Female subject of childbearing potential does not plan pregnancy for at least one year following the index procedure. For a female of childbearing potential, a pregnancy test must be performed with negative results known within seven days prior to index procedure.

Exclusion Criteria:

1. Cardiac Resynchronization Therapy (CRT) or ICD pacing lead placement ≤ 60 days prior to enrollment;
2. Valvular heart disease, which in the opinion of the investigator, will require surgery;
3. Functional Mitral Regurgitation greater than moderate (i.e. EROA>20mm sq.) and primary MR (including MR due to papillary muscle rupture);
4. Need for coronary revascularization, in the opinion of the site investigator;
5. Peak Systolic Pulmonary Arterial Pressure > 60 mm Hg via echo or right heart catheterization and/or evidence of cor pulmonale;
6. Myocardial Infarction within 90 days prior to enrollment;
7. Within the last six months, a prior CVA or TIA, or any intracranial hemorrhage, or any permanent neurologic deficit, or any known intracranial pathology;
8. Co-morbid disease process with life expectancy of less than one year or active malignancy not in remission;
9. Any solid organ transplant or is on waiting list for any solid organ transplant other than cardiac; Page 6 of 64 BioVentrix CIP-0067, Rev A
10. Chronic renal failure with a serum creatinine >2.5 mg/dL and/or GFR<30ml/min;
11. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
12. Presence of significant ventricular arrhythmias
13. Contraindication or inability to adhere to systemic anticoagulation;
14. Known hypersensitivity or contraindication to device materials;
15. Previous pericardiotomy or left thoracotomy;
16. Pathology/previous surgery/radiation therapy of the right neck that would interfere with placement of a 14F delivery catheter;
17. Prior open heart surgery or significant pericarditis;
18. Calcified ventricular wall in the area of intended anchor implants as verified by cardiac imaging;
19. Thrombus or intra-ventricular mass in the left atrium or ventricle as verified by cardiac imaging that has not been adequately treated with anticoagulant.
20. Functioning pacemaker leads in antero-apical RV, which, in the opinion of the investigator, would interfere with anchor placement.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai, New York, NY; Jerry Estep, MD, Principal Investigator — Cleveland Clinic Florida, Weston, FL
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania